CLINICAL TRIAL: NCT02271061
Title: Effects of Elastic Therapeutic Tape on Biomechanical Changes of Knee Joint During Drop Vertical Jump in ACL Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Thammasat University (Other); Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MURA2014/415
Record Dates: First submitted 2014-10-18; First posted 2014-10-22 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kinesio Tape (Experimental): Taping method will be performed in supine position .The taping technique will be started at tibial tuberosity to medial and lateral epicondyles of the femur. The tape will be cut in I shape with 30 cm. The back paper of tape will be removed from the center of tape and both end of the back paper will be placed at each end of tape. Center of the tape will be placed on the tibial tuberosity with no tension. Participants' knee will be bend approximately 20 - 30 degrees. The tape will be pulled at 1/3 of each end with 75% of available tension along the medial and lateral collateral ligaments and the tibia will be pushed to the back. The end of the tape will be placed with no tension toward the medial and lateral aspects of the thigh .
  Interventions: Device: Kinesio tape
- Control tape (Sham Comparator): Apply tape in same technique without tension.
  Interventions: Device: Control tape

INTERVENTIONS:
Device: Kinesio tape — Elastic therapeutic tape is one type of elastic tape that is widely used for various treatment including rehabilitation and sports injuries . The elastic therapeutic tape has different characteristics from other kind of tape. It has ability to stretch around 130 - 140% from original length and recoil back to starting length after applying the tape. Tape produces pulling force on skin which lifts and folds layers of epidermis . Pulling force provides an appropriate alignment which can facilitate and inhibit muscle contraction.It has been claimed for several benefits such as supportingly injured muscles, increased proprioception, stimulated and inhibited muscle activity, relieved pain, increased range of motion, and improved blood and lymph flow.
  Arms: Kinesio Tape
Device: Control tape — Apply tape in same technique without tension.
  Arms: Control tape

SUMMARY:
The purpose of this study to investigate joint angle and joint moment in flexion-extension, adduction-abduction and internal -external rotation of elastic therapeutic tape and elastic therapeutic tape are effective in ACL-injuries subjects during drop vertical jump.This study requires ACL-injuries participants age range between 18 and 45 years old. The 3D motion analysis system (BTS, ITALY) and force plate (Kistler, USA) will be used for measure joint angle and joint moment during drop vertical jump movement.

DETAILED DESCRIPTION:
#Participants ACL-injures subjects ACL-injury group will be recruit people with ACL-injuries with grade I-II at least 8 weeks by measuring joint laxity test by stress X-ray with Telos (side to side difference between 3 - 8 mm.) .

Inclusion criteria of ACL-injuries group are: 1) no collateral ligaments and meniscus injuries , 2) no joint pain and knee joint effusion (less than 2 cm. from the opposite side measuring at joint line, 3) no history of previous injuries in other structure of lower extremities that resulted in ligamentous laxity at ankle and hip, 4) no current medical problems such as vestibular system, visual system or neurological condition that can impair their ability to perform a sidestep cutting task, 5) no joint and structural deformity such as flat feet, genu valgus and genu varus, 6) able to complete functional test (Single hop for distance and Triple hop for distance) which the distance is not less than 85% of unaffected side .

Exclusion criteria included 1) knee joint swelling is greater than 2 cm. of unaffected side, 2) joint laxity test by stress X-ray with Telos (side to side difference greater than 8 mm.)

* Instrumentation

  1. Three-dimensional motion analysis system (Bioengineering Inc., ITALY)
  2. Visual 3D software (C-motion, USA)
  3. A force platform with 60x40x10 centimeters in size (Kistler Instrument Corp., USA)
  4. Running shoes (Adidas) US Size 7 , 8 , 9, 10
  5. Goniometer
  6. Vernier caliber
  7. Measuring tape
  8. Therapeutic tape ; (KinesioTex®)
  9. Telos arthrometer GA III/E (Metax GmbH)
  10. International Knee Documentation Committee Score (IKDC)
  11. Knee Osteoarthritis Outcome Score (KOOS)
* Subject preparation for participants with ACL-injuries Participants will be asked to fill in a questionnaire about age, height, weight and history of injury or musculoskeletal problems. Participants will be informed to make understanding of purposes, methods and advantages of the study. Also, all participants will be asked to sign a consent form. IKDC and KOOD interviews will be conducted.The test including hop test and drop vertical jump will be conducted at Faculty of Medicine Ramathibodi, Mahidol University.

Anthropometric data, navicular drop test, ROM and muscle strength at knee joint will be performed in each participant. Participants will be asked to perform single hop for distance and triple hop on both side of their legs.

Stress X-ray by Telos® Participants will be screened joint laxity by stress x-ray with Telos. Lateral view x-ray will be performed in side lying position with knee flexion between 10 to 20 degrees. Front cushion pad will be applied on distal femur and distal tibia. Pressure load will be applied on 6 cm below knee joint line at 15 daN.

Participants with ACL injuries subjects will rest for 10 minute in the quiet room and elastic therapeutic tape will be applied on affected side. Drop vertical jump will be performed follow by running 30 minutes at speed 7 km/hr. Participants will be asked to perform drop vertical jump task again after running.

Drop vertical jump Drop vertical jump landing trails was performed on 31 cm. box . Participants were informed to jump with two hands over head as high as possible and landing on force plate with each foot on separate force plate . Participants were asked to perform the task until reach three successful trials. Successful trial was defined as participants can land on force plate with each foot on separate force plate without further steps.

#Parameters

Knee joint angle and moment at initial contact and weight acceptance phase

1. Flexion - Extension
2. Adduction - Abduction
3. Internal - External rotation

   * Statistics All data will be presented in mean ± stand error of mean. All the statistical test will be performed by using the SPSS for window version 17 program. The level of significance for difference between groups will be set at p< 0.05.

Comparison of 3D joint angles and moments between affected leg and unaffected leg in ACL-injuries group during side step movement will be tested by Paired T test.

ELIGIBILITY:
Inclusion Criteria:

1. ACL-injuries with grade I-II at least 8 weeks by measuring joint laxity test by stress X-ray with Telos (side to side difference between 3 - 8 mm.)
2. No collateral ligaments and meniscus injuries
3. No joint pain and knee joint effusion (less than 2 cm. from the opposite side measuring at joint line
4. No history of previous injuries in other structure of lower extremities that resulted in ligamentous laxity at ankle and hip
5. No current medical problems such as vestibular system, visual system or neurological condition that can impair their ability to perform a sidestep cutting task
6. No joint and structural deformity such as flat feet, genu valgus and genu varus
7. Able to complete functional test (Single hop for distance and Triple hop for distance) which the distance is not less than 85% of unaffected side

Exclusion Criteria:

1. Knee joint swelling is greater than 2 cm. of unaffected side
2. Joint laxity test by stress X-ray with Telos (side to side difference greater than 8 mm.)
3. Unable to complete functional test (Single hop for distance and Triple hop for distance) which the distance is less than 85% of unaffected side

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Knee joint motion | 6 months
  Knee joint angle and moment at initial contact and weight acceptance phase
  1. Flexion - Extension
  2. Adduction - Abduction
  3. Internal - External rotation

CONTACTS AND LOCATIONS:
Overall Officials: Wat Limruengrangrat, PhD, Principal Investigator — Collage of Sports Sciences and Technology, Mahidol University

REFERENCES:
- [Background] Beldame J, Bertiaux S, Roussignol X, Lefebvre B, Adam JM, Mouilhade F, Dujardin F. Laxity measurements using stress radiography to assess anterior cruciate ligament tears. Orthop Traumatol Surg Res. 2011 Feb;97(1):34-43. doi: 10.1016/j.otsr.2010.08.004. Epub 2010 Dec 18. PMID 21169080
- [Background] Beldame J, Mouchel S, Bertiaux S, Adam JM, Mouilhade F, Roussignol X, Dujardin F. Anterior knee laxity measurement: comparison of passive stress radiographs Telos((R)) and "Lerat", and GNRB((R)) arthrometer. Orthop Traumatol Surg Res. 2012 Nov;98(7):744-50. doi: 10.1016/j.otsr.2012.05.017. Epub 2012 Oct 16. PMID 23084264
- [Background] Bjornaraa J, Di Fabio RP. Knee kinematics following acl reconstruction in females; the effect of vision on performance during a cutting task. Int J Sports Phys Ther. 2011 Dec;6(4):271-84. PMID 22163089
- [Background] Ford KR, Myer GD, Hewett TE. Valgus knee motion during landing in high school female and male basketball players. Med Sci Sports Exerc. 2003 Oct;35(10):1745-50. doi: 10.1249/01.MSS.0000089346.85744.D9. PMID 14523314
- [Background] Hewett TE, Myer GD, Ford KR, Heidt RS Jr, Colosimo AJ, McLean SG, van den Bogert AJ, Paterno MV, Succop P. Biomechanical measures of neuromuscular control and valgus loading of the knee predict anterior cruciate ligament injury risk in female athletes: a prospective study. Am J Sports Med. 2005 Apr;33(4):492-501. doi: 10.1177/0363546504269591. Epub 2005 Feb 8. PMID 15722287
- [Background] McLean SG, Huang X, van den Bogert AJ. Association between lower extremity posture at contact and peak knee valgus moment during sidestepping: implications for ACL injury. Clin Biomech (Bristol). 2005 Oct;20(8):863-70. doi: 10.1016/j.clinbiomech.2005.05.007. PMID 16005555
- [Background] Swirtun LR, Jansson A, Renstrom P. The effects of a functional knee brace during early treatment of patients with a nonoperated acute anterior cruciate ligament tear: a prospective randomized study. Clin J Sport Med. 2005 Sep;15(5):299-304. doi: 10.1097/01.jsm.0000180018.14394.7e. PMID 16162987